CLINICAL TRIAL: NCT00003712
Title: A Phase I Study of the Safety, Tolerability, and Pharmacokinetics of Intravenous CCI-779 Given Once Daily for 5 Days Every 2 Weeks to Patients With Advanced Solid Tumors
Brief Title: CCI-779 in Treating Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: National Cancer Institute (NCI) (NIH); University of Texas (Other); Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000066820; P30CA054174 (NIH); UTHSC-9785011303 (Other: UTHSCSA IRB); SACI-IDD-98-02 (Other: San Antonio Cancer Institute); W-AR-3066K1-100-US (Other: Wyeth); NCI-V98-1506 (Other: NCI)
Record Dates: First submitted 1999-11-01; First posted 2003-07-15 (Estimated); Last update posted 2012-08-09 (Estimated); Status verified 2012-08

CONDITIONS: Brain and Central Nervous System Tumors; Metastatic Cancer; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: recurrent adult brain tumor; unspecified adult solid tumor, protocol specific; tumors metastatic to brain
MeSH Terms: conditions — Central Nervous System Neoplasms; Neoplasm Metastasis; Brain Neoplasms | interventions — temsirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: temsirolimus — •Part I: Patients receive CCI-779 IV over 30 minutes on days 1-5, followed by a 9 day rest period. Treatment courses repeat every 2 weeks in the absence of disease progression or unacceptable toxicity.
  The maximum tolerated dose for part I is defined as the dose level at which 33% of patients experience dose limiting toxicity.
  •Part II: Patients receive the same treatment schedule as part I. Three patients with CNS tumors are entered at the dose of CCI-779 determined to be the MTD in Part I. At least 3 patients are entered at each dose level in part II.

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase I trial to study the effectiveness of CCI-779 in treating patients who have advanced solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the safety, tolerability, and maximum tolerated dose (MTD) of CCI-779 in patients with advanced solid tumors (part I) who are not receiving anticonvulsant therapy.
* Determine the safety, tolerability, and MTD in patients with recurrent gliomas or brain metastases (part II) who are receiving anticonvulsant therapy.
* Determine the preliminary pharmacokinetic profile and antitumor activity of CCI-779 in these patients.

OUTLINE: This is an open-label, dose-escalation study.

* Part I: Patients receive CCI-779 IV over 30 minutes on days 1-5, followed by a 9 day rest period. Treatment courses repeat every 2 weeks in the absence of disease progression or unacceptable toxicity.

The maximum tolerated dose for part I is defined as the dose level at which 33% of patients experience dose limiting toxicity.

* Part II: Patients receive the same treatment schedule as part I. Three patients with CNS tumors are entered at the dose of CCI-779 determined to be the MTD in Part I. At least 3 patients are entered at each dose level in part II.

PROJECTED ACCRUAL: Approximately 20 patients will be accrued for part I for this study within 8 months, and 12 patients will be accrued for part II within 7 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

Part I:

* Histologically proven advanced solid tumors that are refractory or for which no curative therapy exists
* No CNS metastases, peritumoral edema, or symptomatic brain metastases (part I)
* Measurable or evaluable disease

Part II:

* Histologically proven recurrent gliomas or brain metastases for which no curative therapy exists
* Receiving anticonvulsants
* Measurable or evaluable disease

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-2

Life expectancy:

* At least 3 months

Hematopoietic:

* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* Hemoglobin at least 9 g/dL

Hepatic:

* Bilirubin less than 1.5 mg/dL
* AST or ALT less than 3 times upper limit of normal (ULN) (less than 5 times ULN if liver metastases)

Renal:

* Creatinine less than 2 mg/dL

Cardiovascular:

* No unstable angina
* No myocardial infarction within past 6 months
* No maintenance therapy for life-threatening arrhythmias

Other:

* Not pregnant or nursing
* Fertile patients must use effective contraception
* HIV negative
* No active infection or other serious concurrent illness
* Triglycerides no greater than 300 mg/dL
* Cholesterol no greater than 350 mg/dL
* No known hypersensitivity to macrolide antibiotics (e.g., clarithromycin, erythromycin, or azithromycin)

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* At least 3 weeks since prior chemotherapy (6 weeks since nitrosoureas and mitomycin)
* No other concurrent chemotherapy

Endocrine therapy:

* Concurrent corticosteroids used to reduce edema in patients with primary or metastatic CNS tumors allowed
* No concurrent hormonal therapy

Radiotherapy:

* At least 3 weeks since prior radiotherapy
* No concurrent radiotherapy

Surgery:

* Not specified

Other:

* At least 1 month since prior investigational agents
* At least 3 weeks since prior immunosuppressive therapy
* No concurrent anticonvulsant therapy (part I)
* No concurrent immunosuppressive therapy (e.g., terfenadine, cisapride, astemizole, pimozide)
* No known agents that inhibit or induce cytochrome p450

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2001-01; Primary Completion 2002-06 (Actual); Study Completion 2002-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric K. Rowinsky, MD, Study Chair — San Antonio Cancer Institute
Locations (2):
- United States (2):
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - San Antonio Cancer Institute, San Antonio, Texas